CLINICAL TRIAL: NCT01761747
Title: Phase II Study of Ponatinib in Advanced Lung and Head and Neck Cancers With FGFR Kinase Alterations
Brief Title: Ponatinib for Squamous Cell Lung and Head and Neck Cancers
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: FDA hold and toxicity associated with study drug
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Peter S. Hammerman, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-327
Record Dates: First submitted 2012-09-26; First posted 2013-01-07 (Estimated); Results first posted 2014-12-23 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Non-Small Cell Lung Cancer, Head and Neck Cancer
Keywords: Squamous Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Head and Neck Neoplasms; Carcinoma, Squamous Cell | interventions — ponatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ponatinib Treatment Arm (Experimental): Ponatinib taken by mouth daily
  Interventions: Drug: ponatinib

INTERVENTIONS:
Drug: ponatinib
  Other Names: AP24534

SUMMARY:
This research study is a Phase II clinical trial, which tests the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific cancer. "Investigational" means that the drug is being studied. It also means that the FDA has not yet approved ponatinib for use in patients, including people with your type of cancer.

In order to participate on this study, it must first be determined whether or not a patient's lung or head and neck squamous cell cancer (SCC) has an alteration in FGFR kinase is made from an experimental test on your squamous cell cancer tissue sample. This experimental test is a "genetic test" or "genotyping test", which is a method used to study a tumor's genes. The results are for research purposes only and are not considered "genetic testing" for the purpose of diagnosing medical conditions. Cancers develop as a result of changes that occur in human genetic material (DNA); these changes are called mutations or alterations. This experimental test gives no information about any of the genes in the normal cells of the patient's body, but it helps identify abnormal genes (like FGFR kinase mutations or alterations) usually found only in cancer cells. We will use this experimental test to determine whether or not a tumor contains a required alteration/mutation and thus may respond to ponatinib.

Ponatinib is an investigational, oral anti-cancer drug designed to inhibit abnormal proteins found in cancer cells and may cause those cancer cells to die. In laboratory testing, ponatinib has been shown to inhibit a family of proteins called FGFR kinases, and this genetic alteration/mutation has been found in some squamous cell lung cancers. There is laboratory evidence that alterations/mutations in FGFR kinases in squamous cell lung cancers may be driving the growth of these tumors and that inhibiting these FGFR kinases with ponatinib may decrease or stop the growth of lung SCC.

In this research study, we are looking to see if the study drug, ponatinib, can keep cancer from growing.

DETAILED DESCRIPTION:
Patients will be asked to undergo some screening tests or procedures to find out if they can be in the research study. Many of these tests and procedures are likely to be part of regular cancer care and may be done even if it turns out that an individual does not take part in the research study. If a patient has had some of these tests or procedures recently, they may or may not have to be repeated. These screening tests include: medical history, physical examination, vital signs, performance status, assessment of tumor(s), CT scan or MRI scan of brain, routine blood tests, urine pregnancy test for women of childbearing potential and electrocardiogram. Additionally at the time of screening patients will undergo collection of an archival tumor tissue sample for tumor mutation testing.

If a patient takes part in this research study, he or she will be given a study drug-dosing calendar for each treatment cycle. Each treatment cycle lasts 4 weeks during which time the patient will be taking the study drug by mouth daily. The number of cycles the patient will receive will depend on how the patient is tolerating the ponatinib and if your cancer has worsened.

There is a possibility that the following tests or procedures may need to be done at times other than those listed below. These may be done if the research doctors determine they are medically necessary to monitor illness or any side effects a patient may be experiencing. It is important that patients call their research doctor if at any time they are experiencing side effects they cannot tolerate.

During all cycles patients will have a physical exam and be asked questions about their general health and specific questions about any problems that they might be having and any medications they might be taking.

If the patient's disease progresses while you are on this study, they will be given the option of consenting to a new biopsy for research purposes at no financial cost to the patient.

The investigators would like to keep track of your medical condition for the rest of each patient's life. The investigators would like to do this by calling every six months to see how the patients are doing. Keeping in touch with checking their condition helps the investigators look at the long-term effects of the research study.

ELIGIBILITY:
Inclusion Criteria:

* Measurable disease
* Documented evidence of disease progression following most recent therapy
* Estimated life expectancy greater than 12 weeks

Exclusion Criteria:

* Pregnant or breastfeeding
* Prior chemotherapy or brain radiotherapy within 4 weeks of entering study
* Receiving other investigational agents
* Untreated or progressive brain metastases
* Prior treatment with or allergic reactions attributed to compounds of similar chemical or biologic composition to ponatinib
* Known HIV positive on combination antiretroviral therapy
* Clinically uncontrolled hypertension
* Previous or concurrent malignancy except adequately treated basal or squamous cell skin cancer, in situ carcinoma of the cervix, or other solid tumor treated curatively and without evidence of recurrence for at least 5 years
* Active or uncontrolled clinically significant infection
* Chronic GI disease that may affect bioavailability of ponatinib
* History of significant bleeding disorder unrelated to cancer
* Uncontrolled intercurrent illness
* Clinically significant ventricular arrythmia
* History of chronic pancreatitis, alcohol abuse or uncontrolled hypertriglyceridemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hammerman, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Groups:
- Ponatinib Treatment Arm: Ponatinib taken by mouth daily
  ponatinib
Period: Overall Study
Arm/Group | Ponatinib Treatment Arm
Started | 3
Completed | 2
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ponatinib Treatment Arm
Number analyzed (Participants) | 3
Age, Continuous [Mean (Full Range); unit: years] | 61 [37 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 3
Region of Enrollment [Number; unit: participants]
  United States | 3
Disease [Number; unit: participants] — Non-small cell lung cancer
  participants | 3

OUTCOME MEASURES:

1. Primary Outcome: Response Rate of Patients With Lung or Head and Neck SCC Treated With Ponatinib
Description: Investigate the response rate of patients with previously treated lung or head and neck SCC to ponatinib as defined by the proportion of subjects with investigator-assessed confirmed complete response (CR) or partial response (PR).
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR."
Time Frame: 2 years
Measure: Number; unit: percentage of subjects with response
Arm/Group | Ponatinib Treatment Arm
Number analyzed (Participants) | 3
percentage of subjects with response | 0

2. Secondary Outcome: Prevalence of Specific FGFR Amplifications/Mutations in the Study Population
Description: Test tumor DNA using molecular assays to measure the frequency of FGFR amplifications and mutations in study patients
Time Frame: 2 years
Population: 2 participants had FGFR amplification, one with FGFR mutation
Measure: Number; unit: participants
Arm/Group | Ponatinib Treatment Arm
Number analyzed (Participants) | 3
participants | 3

3. Secondary Outcome: Progression-free Survival
Description: Establish the progression-free survival of patients with SCC treated with ponatinib as defined by time to development of progression by RECIST criteria.
Time Frame: 2 years
Measure: Mean (Full Range); unit: days
Arm/Group | Ponatinib Treatment Arm
Number analyzed (Participants) | 2
days | 44 [32 to 55]

4. Secondary Outcome: Define Toxicities of Ponatinib
Description: Number of Participants with Adverse Events as a Measure of Safety and Tolerability
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Ponatinib Treatment Arm
Number analyzed (Participants) | 3
participants | 2

5. Secondary Outcome: Overall Survival
Description: Measure the overall survival time of patients treated with ponatinib
Time Frame: 2 years
Measure: Mean (Full Range); unit: days
Arm/Group | Ponatinib Treatment Arm
Number analyzed (Participants) | 3
days | 276 [48 to 588]

6. Secondary Outcome: Disease Control
Description: Measure the disease control rate of patients treated with ponatinib
Time Frame: 2 years
Measure: Number; unit: percentage of subjects
Arm/Group | Ponatinib Treatment Arm
Number analyzed (Participants) | 2
percentage of subjects | 0

7. Secondary Outcome: Determine the Correlation FGFR Amplifications/Mutations With Patient Age, Sex, Disease Stage, Prior Response to Treatment and Smoking History
Description: For subjects with FGFR amplifications and for FGFR mutations we will ascertain the age, sex, disease stage, prior response to treatment and smoking history from past medical records and measure whether there are differences in these variables among subjects with amplification versus mutation.
Time Frame: 2 years
Population: Too few subjects were enrolled on study to permit this outcome measure analysis.
Arm/Group | Ponatinib Treatment Arm
Number analyzed (Participants) | 0

8. Secondary Outcome: Define the Response Rate to Ponatinib is Patients With FGFR Amplifications Versus Mutations
Description: Identify the response rate to ponatinib for FGFR specific FGFR amplifications/mutations.
Time Frame: 2 years
Population: There were no observed responses on study so this outcome could not be determined.
Arm/Group | Ponatinib Treatment Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: One individual withdrew consent the day after enrolling on study and was not dosed. Therefore only two individuals were evaluable for treatment-related toxicities.
Arm/Group | Ponatinib Treatment Arm
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ponatinib Treatment Arm (N=2)
Pancreatits (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ponatinib Treatment Arm (N=2)
Fatigue (General disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Mucositis (Gastrointestinal disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neuropathy (Nervous system disorders) | 1
Hepatitis (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No